CLINICAL TRIAL: NCT01179542
Title: The Involvement of Eukaryotic Translation Initiation Factor 4E (eIF4E) in Human Placental Implantation and in the Pathological Pregnancies: Preeclampsia and IUGR.
Status: Withdrawn | Type: Observational
Why Stopped: recruiting problems
Sponsor: Meir Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: mmc10134-2010ctil
Record Dates: First submitted 2010-08-10; First posted 2010-08-11 (Estimated); Last update posted 2017-09-13 (Actual); Status verified 2010-08

CONDITIONS: Pregnancy; Preeclampsia
Keywords: iugr pet eIF4E Translation Initiation Factor; 4E (eIF4E) in Human Placental Implantation and in the Pathological Pregnancies: Preeclampsia and IUGR
MeSH Terms: conditions — Pre-Eclampsia; Fetal Growth Retardation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- first trimester: first trimester
- third trimester: third trimester
- prgnancies complicated with IUGR: prgnancies complicated with IUGR
- preeclampsia: preeclampsia

SUMMARY:
The involvement of eukaryotic translation initiation factor 4E (eIF4E) in human placental implantation and in the pathological pregnancies: preeclampsia and IUGR.

DETAILED DESCRIPTION:
4 groups

ELIGIBILITY:
Inclusion Criteria:

* post TOP or DELIVERY

Exclusion Criteria:

-

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Only the Placenta aftr delivery or abortion
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2010-09; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
measure the Translation Initiation effect of experimental variables observational studies | 2 years